CLINICAL TRIAL: NCT04018599
Title: A Phase I, Randomized, Open-label, Parallel-group Study to Determine the Pharmacokinetics, Safety, and Tolerability of MSB11022 (Proposed Adalimumab Biosimilar) Following a Single Subcutaneous Injection by an Auto-injector or by a Pre-filled Syringe in Healthy Subjects
Brief Title: Comparison of PK and Tolerability of MSB11022 Administered by AI or PFS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fresenius Kabi SwissBioSim GmbH (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FKS022-001
Record Dates: First submitted 2019-07-11; First posted 2019-07-12 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis; Polyarticular Juvenile Idiopathic Arthritis; Psoriatic Arthritis; Ankylosing Spondylitis; Crohn Disease; Ulcerative Colitis; Plaque Psoriasis; Pediatric Plaque Psoriasis; Pediatric Crohns Disease; Hidradenitis Suppurativa; Non-infectious Uveitis
Keywords: Biosimilar; Adalimumab; MSB11022
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Juvenile; Arthritis, Psoriatic; Spondylitis, Ankylosing; Crohn Disease; Colitis, Ulcerative; Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 40 mg MSB11022 via Auto-injector (Experimental): Participants will receive a single dose of 40 mg/0.8 mL of MSB11022 via an auto-injector on Day 1.
  Interventions: Drug: 40 mg MSB11022
- 40 mg MSB11022 via Pre-filled Syringe (Experimental): Participants will receive a single dose of 40 mg/0.8 mL of MSB11022 via a pre-filled syringe on Day 1.
  Interventions: Drug: 40 mg MSB11022

INTERVENTIONS:
Drug: 40 mg MSB11022 — Single dose, as a solution, administered subcutaneously, using an auto-injector.
  Arms: 40 mg MSB11022 via Auto-injector
Drug: 40 mg MSB11022 — Single dose, as a solution, administered subcutaneously, using a pre-filled syringe.
  Arms: 40 mg MSB11022 via Pre-filled Syringe

SUMMARY:
The primary objective of this study is to demonstrate equivalence of the pharmacokinetic (PK) profile of MSB11022 administered by either an auto-injector (AI) or a pre-filled syringe (PFS) as single subcutaneous (s.c.) injection of 40 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign the informed consent form (ICF).
2. Healthy male subjects and female subjects of non-childbearing and childbearing potential.
3. Aged 18 to 55 years, inclusive, at screening.
4. Have all screening results (vital signs, physical examination, clinical laboratory tests, 12-lead ECG) within the normal range or outside the normal range but assessed as not clinically significant by the Investigator.
5. Body weight between 50.0 and 100.0 kg, inclusive, and a body mass index between 18.5 and 30.0 kg/m2, inclusive.
6. Male subjects must be either surgically sterile or willing to use contraceptive methods until 5 months after the dose of investigational medicinal product (IMP).
7. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and before randomization. WOCBP must agree to use highly effective methods of contraception to prevent pregnancy for at least 4 weeks before randomization until 5 months after the dose of IMP. For all postmenopausal female subjects, serum follicle-stimulating hormone (FSH) is tested at screening to identify their postmenopausal status.
8. Willing and able to comply with scheduled visits, treatment plan, laboratory tests and all other study procedures.

Exclusion Criteria:

1. Female subjects must not be pregnant or lactating at screening through at least 5 months after the last treatment with IMP.
2. A history and/or current presence of clinically significant atopic allergy (eg, asthma including childhood asthma), hypersensitivity or allergic reactions (either spontaneous or following drug administration), including known or suspected clinically relevant drug hypersensitivity to any components of the study drug formulations, comparable drugs, or to latex. Mild hay fever is allowed if outside of acute exacerbation requiring treatment. Assessment of clinical significance of reported atopic or allergic condition in medical history of participant is at Investigator decision.
3. Have either active or latent tuberculosis (TB) as indicated by a positive QuantiFERON®-TB Gold test or have a history of TB. Subjects who have an indeterminate QuantiFERON-TB Gold test result may be re-tested once during screening. If the re-test result is negative, the subject is eligible to participate in the study. If the re-test result is indeterminate again or positive, the subject is NOT eligible to participate in the study.
4. Lifetime history of invasive systemic fungal infections (eg, histoplasmosis) or other opportunistic infections, including recurrent or chronic local fungal infections.
5. Have had a serious infection (associated with hospitalization and/or which required intravenous anti-infectives or intravenous antibiotics) within 6 months prior to study drug administration and/or a significant infection (excluding resolved infections like a mild common cold) within 2 weeks prior to the screening or during the screening period unless the infection has resolved completely within 2 weeks before admission.
6. Have had herpes zoster

   1. within the last year, or
   2. more than 2 herpes zoster infections in their lifetime prior to randomization.
7. History or presence (at time of screening or randomization) of frequent (ie, requiring treatment more than 3 times a year), chronic or recurrent infections.
8. Have previously been exposed to adalimumab or approved or proposed adalimumab biosimilar drugs if known. Have been exposed to any anti-tumor necrosis factor alfa class drug whether approved drug or investigational drug\proposed biosimilar.
9. Intake of an investigational drug in another study within 3 months or 5 half-lives, whichever is longer, before the intake of the IMP in this study or planned intake of an investigational drug during the course of this study.
10. Use of depot injectable solutions (except for depot contraception drugs) within 6 months before randomization.
11. Smoking more than equivalent of (as determined by investigator) 10 cigarettes per day and/or inability to refrain from smoking or consuming nicotine containing products during the residential stay at the trial site.
12. History of alcohol abuse within one year from screening and/or inability to refrain from intake of alcoholic beverages from 48 hours prior to Day -1 until Day 14 postdose or a positive screen for alcohol on admission to the clinical site prior to study drug administration.
13. Positive screen for drugs of abuse at screening or at admission to the clinical site prior to study drug administration.
14. Donated more than 450 mL of blood within 60 days or 450 mL of blood products (eg, plasma, platelets) within 2 weeks prior to admission to the clinical site or intend to donate during the study.
15. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), dietary supplements or herbal medication during the 2 weeks prior to study drug administration or longer if the medication has a long half-life. For female subjects, oral contraceptives and hormone replacement therapy are allowed.
16. History of cancer including lymphoma, leukemia, and skin cancer.
17. Impaired liver function as determined at screening or admission to the clinic by one of the following:

    * Serum alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 times the upper limit of normal (ULN) at screening or admission to the clinic.
    * A positive hepatitis C virus (HCV) antibody test or hepatitis B surface antigen (HBsAg) test and/or core antibody test for immunoglobulin G (IgG) and/or immunoglobulin M (IgM) at screening.
18. History of or current signs or symptoms of demyelinating disease including optic neuritis and/or multiple sclerosis.
19. History of immunodeficiency (including a positive test for human immunodeficiency virus [HIV] 1 or 2 antibodies) or other clinically significant immunological disorders, or autoimmune disorders, (eg, rheumatoid arthritis, lupus erythematosus, scleroderma).
20. History of and/or current gastrointestinal, renal, cardiovascular, hematological (including pancytopenia, aplastic anemia or blood dyscrasia), metabolic (including known diabetes mellitus), central nervous system or pulmonary disease considered as significant by the Investigator.
21. Received a live vaccine within 12 weeks prior to screening visit or plan for any such vaccination during the study or within 4 months after study drug administration.
22. Any abnormal skin conditions or potentially obscuring tattoos, pigmentation, or lesions in the areas intended for s.c. injection, that in opinion of Investigator do not allow assessment of local tolerability.
23. Legal incapacity or limited legal capacity.
24. Significant concurrent disease or a known medical condition which would make the participant unfit to participate in the study as per Investigator assessment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve from Time Zero to Infinity (AUC0-inf) for MSB11022 | Pre-dose (-1 hour), 4, 8, 12, 24, 48, 72, 96, 120,144,168, 192, 240, 336, 504, 672, 840,1008, 1344 and 1680 hours post-dose
Maximum Observed Plasma Concentration (Cmax) for MSB11022 | Pre-dose (-1 hour), 4, 8, 12, 24, 48, 72, 96, 120,144,168, 192, 240, 336, 504, 672, 840,1008, 1344 and 1680 hours post-dose
Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-last) for MSB11022 | Pre-dose (-1 hour), 4, 8, 12, 24, 48, 72, 96, 120,144,168, 192, 240, 336, 504, 672, 840,1008, 1344 and 1680 hours post-dose

SECONDARY OUTCOMES:
Time to Reach the Maximum Plasma Concentration (Tmax) for MSB11022 | Pre-dose (-1 hour), 4, 8, 12, 24, 48, 72, 96, 120,144,168, 192, 240, 336, 504, 672, 840,1008, 1344 and 1680 hours post-dose
Terminal Rate Constant (λz) for MSB11022 | Pre-dose (-1 hour), 4, 8, 12, 24, 48, 72, 96, 120,144,168, 192, 240, 336, 504, 672, 840,1008, 1344 and 1680 hours post-dose
Terminal Half-life (t1/2) for MSB11022 | Pre-dose (-1 hour), 4, 8, 12, 24, 48, 72, 96, 120,144,168, 192, 240, 336, 504, 672, 840,1008, 1344 and 1680 hours post-dose
Apparent Total Clearance (CL/F) for MSB11022 | Pre-dose (-1 hour), 4, 8, 12, 24, 48, 72, 96, 120,144,168, 192, 240, 336, 504, 672, 840,1008, 1344 and 1680 hours post-dose
Number of Participants with at Least One Treatment-Emergent Adverse Event (TEAE) | Day 1 (post-dose) to Day 71
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. TEAEs are defined as undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment AE. A TEAE is an AE that occurs only once treatment has started.
Number of Participants with at Least One Serious Adverse Event (SAE) | Screening (up to 28 days prior to study admission) to Day 71
  An SAE is defined as an AE occurring during any study phase that fulfills one or more of the following criteria:
  * Results in death.
  * Requires hospitalization (in-patient treatment) or prolongation of existing hospitalization.
  * Is life-threatening.
  * Results in persistent or significant disability or incapacity.
  * Is a congenital anomaly or birth defect.
  * Is otherwise considered to be medically important.
Number of Participants with at Least One Adverse Event of Special Interest (AESI) | Screening (up to 28 days prior to study admission) to Day 71
  An AESI is defined as a hypersensitivity reaction of Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or above.
Number of Participants with an Injection Site Reaction (ISR) | Day 1 (post-dose) to Day 71
  Local tolerability will be assessed be evaluating the site of administration. The investigator or designee will check for the presence of injection site reactions, including, erythema, rash, tenderness, swelling, itching, bruising, or other abnormalities.
Number of Participants who Experience a Clinically Significant Change in Vital Sign Results | Screening (up to 28 days prior to study admission) to Day 71
  Vital sign measurements will include Systolic and diastolic blood pressure, pulse, body temperature and respiratory rate.
Number of Participants who Experience a Clinically Significant Change in Clinical Laboratory Results | Screening (up to 28 days prior to study admission) to Day 71
  Parameters will include clinical chemistry, coagulation, hematology, urinalysis and serology.
Number of Participants who Experience a Clinically Significant Change in Electrocardiogram (ECG) Results | Screening (up to 28 days prior to study admission) to Day 71
  A standard 12-lead ECG will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Radmila Kanceva, MD, PhD, Study Director — Fresenius Kabi SwissBioSim GmbH
Locations (2):
- United States (2):
  - PRA Health Sciences (PRA) - Early Development Services (EDS), Lenexa, Kansas
  - PRA-EDS, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sabet A, Dickerson DS, Kunina EE, Buccarello AL, Monnet J. A Randomised Controlled Trial Comparing the Pharmacokinetics and Tolerability of the Proposed Adalimumab Biosimilar MSB11022 Delivered via Autoinjector and Pre-filled Syringe in Healthy Subjects. Rheumatol Ther. 2022 Apr;9(2):693-704. doi: 10.1007/s40744-022-00432-1. Epub 2022 Mar 9. PMID 35262901